CLINICAL TRIAL: NCT02814201
Title: Study of Motor Slowing in Parkinson's Disease by a Computerized Mental Chronometry Paradigm
Acronym: ERAMPPCI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI10-DR-DURU
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson Disease; Huntington Disease
Keywords: Motor slowing; Computerized mental chronometry paradigm
MeSH Terms: conditions — Parkinson Disease; Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Parkinson best-On: two hours after taking two tablets of 125 mg dispersible Modopar®
  Interventions: Behavioral: SRT
- Parkinson worst-off: after a drug withdrawal period ( morning fasting all dopaminergic treatment since the day before midnight)
  Interventions: Behavioral: SRT
- Huntington
  Interventions: Behavioral: SRT
- Control: Data collected from the existing database
  Interventions: Behavioral: SRT

INTERVENTIONS:
Behavioral: SRT — simple reaction time ( SRT) defined as the fastest response time to a target stimulus ( phase "worst -off" at the Parkinson's patient )

SUMMARY:
Action slowing has been demonstrated in many diseases. Parkinson's disease (PD) and Huntington's disease (HD) are two neurodegenerative diseases affecting the basal ganglia, particularly the medial globus pallidus, and the clinical expression of these two diseases is characterized by a combination of motor and cognitive disorders, but with two opposing patterns of dysfunction. Action slowing has been demonstrated in both of these diseases and has been extensively studied in Parkinson's disease, suggesting a perceptive-cognitive origin. Far fewer studies have been conducted in Huntington's disease. However, all of these studies were performed with different methodologies in small cohorts and the value of the proposed study is to use a validated and standardized computerized mental chronometry paradigm, providing a better understanding of the mechanisms of action slowing in these two diseases and to more clearly define a disease-specific profile.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* French mother tongue
* MMSE > 20/30
* Specific to the MP and MH:

  * Parkinson's disease:

    * defined by the criteria of the UKPDSBB
    * stage 1 , 2 or 3 Hoehn and Yahr (ON)
    * age of onset of the disease known
    * brain MRI performed during follow-up
  * Huntington disease :

    * genetically defined (CAG > 35)
    * weaning neuroleptic ( Tercian® and Solian® : 2 days; Haldol® : 5 days ; Tiapridal® and Xenazine : 1 day ; Zyprexa® : 4 days)
    * Early stage : Fahn and Shoulson I and II is a CFT score between 7 and 13

Exclusion Criteria:

* Illiteracy, writing or reading difficulties
* Visual perceptual auditory deficit or preventing reading, drawing, writing or understanding instructions
* Visual hallucinations
* Significant history may sound on cognition (unbalanced thyroid dysfunction, ischemic heart disease or embolic unstabilized or symptomatic, progressive neoplasia, chronic alcoholism weaned or not)
* Current or previous neurological diseases other than MH or MP: ischemic cerebral vascular accident or bleeding, head injuries (loss of higher knowledge in 15 minutes), epilepsy requiring treatment.
* Psychiatric disorders depression unless treated (stable treatment for 1 month)
* Psychotropic treatment (except anxiolytic, antidepressant steady since 1 month)
* Inability to achieve an autonomous operation without technical assistance over a distance of 20 meters.
* Inability to stand without technical assistance for 30 seconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hoehn and Yahr stage 1 to 3 Parkinson's disease and patients with Shoulson stage I and II Huntington's disease, in whom admission to the Neurology ward is scheduled in the context of their follow-up, comprising a neuropsychological assessment (together with an acute L-dopa administration test for Parkinsonian patients) will be included
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
SRT | Day 0
  simple reaction time ( SRT) defined as the fastest response time to a target stimulus ( phase "worst -off" at the Parkinson's patient )

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KRYSTKOWIAK, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France